CLINICAL TRIAL: NCT07381673
Title: The Effect of Parental Self-Efficacy for Child Autonomy on Postoperative Pain in Children Undergoing Minor Surgery
Brief Title: Parental Self-Efficacy for Child Autonomy and Postoperative Pain in Children Undergoing Minor Surgery
Acronym: PSE-PAIN-MS
Status: Recruiting | Type: Observational
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Assistant Professor, Agri Ibrahim Cecen University
Other Study IDs: AICU-MS-PAIN-2026
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain
Keywords: Parental Self-Efficacy; Child Autonomy; Postoperative Pain; Minor Surgery; Pediatric Nursing; Family-Centered Care
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children Undergoing Minor Surgery: This cohort includes children aged 3 to 18 years undergoing minor surgical procedures and their parents. Participants are observed prospectively to assess parental self-efficacy for supporting child autonomy and children's postoperative pain levels. No intervention beyond routine clinical care is applied.

SUMMARY:
This study aims to examine the relationship between parental self-efficacy in supporting child autonomy and postoperative pain levels in children undergoing minor surgical procedures. The study will be conducted with children aged 3 to 18 years and their parents at a single hospital in Turkey.Participation in the study is voluntary. Parents will be asked to complete questionnaires assessing their confidence in supporting their child's autonomy during the surgical process. Children's postoperative pain levels will be assessed using an age-appropriate pain rating scale during the early postoperative period.No experimental treatment or additional medical procedures will be performed as part of this study. All data will be collected as part of routine care and questionnaire assessments. The results of this study are expected to contribute to improved family-centered perioperative care for children undergoing minor surgery.

DETAILED DESCRIPTION:
This prospective observational study is designed to investigate the relationship between parental self-efficacy for supporting child autonomy and postoperative pain levels in children undergoing minor surgical procedures.

The study population consists of children aged 3 to 18 years who are scheduled for minor surgery and their parents or legal guardians. Data will be collected at a single tertiary-level state hospital in Turkey. Participation is based on voluntary informed consent obtained from parents, and age-appropriate assent will be obtained from children when applicable.

Parental self-efficacy related to supporting child autonomy during the surgical process will be assessed preoperatively using the Parental Self-Efficacy Scale for Child Autonomy Toward Minor Surgery, a validated questionnaire. Postoperative pain intensity in children will be assessed during the early postoperative period using the Wong-Baker FACES Pain Rating Scale at predefined time points.

No interventions beyond standard clinical care will be implemented as part of the study. The study does not involve the use of investigational drugs, devices, or experimental procedures. All clinical care, including pain management, will be provided according to routine hospital protocols.

Descriptive statistics will be used to summarize participant characteristics and scale scores. The relationship between parental self-efficacy and postoperative pain levels will be analyzed using appropriate correlational and regression-based statistical methods. The findings are expected to support the development of family-centered perioperative nursing approaches aimed at improving postoperative pain outcomes in children undergoing minor surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 18 years
* Scheduled for minor surgical procedures
* Able to understand and respond to age-appropriate pain assessment tools
* Parents or legal guardians able to read and understand Turkish
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Presence of chronic pain conditions
* Neurological or cognitive disorders that may interfere with pain assessment
* Requirement for postoperative intensive care
* Incomplete completion of data collection forms

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of children aged 3 to 18 years undergoing minor surgical procedures and their parents or legal guardians at a single state hospital in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Level | At 0, 2, and 6 hours after surgery
  Postoperative pain intensity measured using the Wong-Baker FACES Pain Rating Scale, scored from 0 (no pain) to 10 (severe pain). Pain assessments will be conducted at multiple predefined time points during the early postoperative period.

SECONDARY OUTCOMES:
Parental Self-Efficacy for Child Autonomy | Preoperative period, prior to surgery
  Parental self-efficacy assessed using the Parental Self-Efficacy Scale for Child Autonomy Toward Minor Surgery, an 18-item Likert-type scale with scores ranging from 1 to 4, where higher total scores indicate higher parental self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan GOKMEN, Doctorate, Principal Investigator — Agri ibrahim Cecen Univercity
Locations (1):
- Dogubayazit State Hospital, Ağrı, Dogubeyazit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves a pediatric population and includes sensitive health-related information collected from children and their parents. Data are collected solely for the purposes defined in the approved study protocol, and sharing individual-level data could compromise participant confidentiality and privacy.

REFERENCES:
- [Background] Pölkki T, Pietilä AM, Vehviläinen-Julkunen K, Laukkala H, Ryhänen P. Parental views on participation in their child's pain relief measures and recommendations to health care providers. Journal of Pediatric Nursing. 2002;17(4):270-278.
- [Background] Semerci R, Ünver S, Topçu SY, Turan FN, Kostak MA, Fındık ÜY. Adaptation of Parental Self-Efficacy Scale for Child Autonomy Toward Minor Surgery to Turkish. Journal of PeriAnesthesia Nursing. 2022;37(5):632-639.
- [Background] Calcaterra V, Ostuni S, Bonomelli I, et al. Music benefits on postoperative distress and pain in pediatric day care surgery. Pediatric Reports. 2014;6(3):5534. doi:10.4081/pr.2014.5534.
- [Background] Cai Y, Lopata L, Roh A, et al. Factors influencing postoperative pain following discharge in pediatric ambulatory surgery patients. Journal of Clinical Anesthesia. 2017;39:100-104.